CLINICAL TRIAL: NCT04738123
Title: A Phase 3, Randomized, Double-blind, Parallel-group, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of KarXT in Acutely Psychotic Hospitalized Adults With DSM-5 Schizophrenia
Brief Title: A Study to Assess Efficacy and Safety of KarXT in Acutely Psychotic Hospitalized Adult Patients With Schizophrenia (EMERGENT-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAR-009
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia; Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline and Trospium Chloride Capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride Capsules — Oral xanomeline 50 mg/trospium 20 mg BID on days 1-2 followed by xanomeline 100 mg/trospium 20 mg BID on days 3-7. The dose is increased to xanomeline 125 mg/trospium 30 mg BID on days 8-35 unless the subject is experiencing adverse events from the xanomeline 100 mg/ trospium 20 mg dose. Subjects who were increased to xanomeline 125 mg/trospium 30 mg will have the option to return to xanomeline 100 mg/ trospium 20 mg depending on clinical response and tolerability.
  Arms: KarXT
Drug: Placebo — Placebo Capsules
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, parallel-group, placebo-controlled, multicenter inpatient study to examine the efficacy and safety of KarXT in adult subjects who are acutely psychotic with a Diagnostic and Statistical Manual Fifth Edition (DSM-5) diagnosis of schizophrenia. The primary objective of the study is to assess the efficacy of KarXT (a fixed combination of xanomeline 125 mg and trospium chloride 30 mg twice daily [BID]) versus placebo in reducing Positive and Negative Syndrome Scale (PANSS) total scores in adult inpatients with a DSM-5 diagnosis of schizophrenia. The secondary objectives of the study are to evaluate improvement in disease severity and symptoms, safety and tolerability, and pharmacokinetics in adult inpatients with a DSM-5 diagnosis of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 to 65 years, inclusive, at screening.
2. Subject is capable of providing informed consent.

   1. A signed informed consent form must be provided before any study assessments are performed.
   2. Subject must be fluent (oral and written) in English or local language to consent
3. Subject has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM-5 criteria and confirmed by Mini International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorder Studies (MINI) version 7.0.2.
4. Subject is experiencing an acute exacerbation or relapse of psychotic symptoms, with onset less than 2 months before screening.

   1. The subject requires hospitalization for this acute exacerbation or relapse of psychotic symptoms.
   2. If already an inpatient at screening, has been hospitalized for less than 2 weeks for the current exacerbation at the time of screening.
5. Positive and Negative Syndrome Scale total score between 80 and 120, inclusive. Score of ≥4 (moderate or greater) for ≥2 of the following Positive Scale (P) items:

   1. Item 1 (P1; delusions)
   2. Item 2 (P2; conceptual disorganization)
   3. Item 3 (P3; hallucinatory behavior)
   4. Item 6 (P6; suspiciousness/persecution)
6. Subjects with no change (improvement) in PANSS total score between screening and baseline (Day -1) of more than 20%.
7. Subject has a CGI-S score of ≥4 at screening and baseline (Day -1) visits.
8. Subject will have been off lithium therapy for at least 2 weeks before baseline and free of all oral antipsychotic medications for at least 5 half-lives or 1 week, whichever is longer, before baseline (Day -1).
9. Subjects taking a long-acting injectable antipsychotic could not have received a dose of medication for at least 12 weeks (24 weeks for INVEGA TRINZA) before baseline visit (Day -1).
10. Subject is willing and able to be confined to an inpatient setting for the study duration, follow instructions, and comply with the protocol requirements.
11. BMI must be ≥18 and ≤40 kg/m2.
12. Subject resides in a stable living situation and is anticipated to return to that same stable living situation after discharge, in the opinion of the investigator.
13. Subject has an identified reliable informant/caregiver.
14. Women of childbearing potential, or men with sexual partners of childbearing potential, must be able and willing to use at least 1 highly effective method of contraception during the study and for 30 days after the last dose of study drug. Sperm donation is not allowed for 30 days after the final dose of study drug.

Exclusion Criteria:

1. Any primary DSM-5 disorder other than schizophrenia within 12 months before screening (confirmed using MINI version 7.0.2 at screening). Symptoms of mild mood dysphoria or anxiety are allowed as long as these symptoms are not the primary focus of treatment. A screening subject with mild substance abuse disorder within the 12 months before screening must be discussed and agreed upon with the medical monitor before they can be allowed into the study.
2. Subjects who are newly diagnosed or are experiencing their first treated episode of schizophrenia.
3. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results.
4. Subjects with HIV, cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections based on either medical history or liver function test results.
5. History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma.
6. History of irritable bowel syndrome (with or without constipation) or serious constipation requiring treatment within the last 6 months.
7. Risk for suicidal behavior during the study as determined by the investigator's clinical assessment and Columbia-Suicide Severity Rating Scale (C-SSRS).
8. Clinically significant abnormal finding on the physical examination, medical history, ECG, or clinical laboratory results at screening.
9. Subjects cannot currently (within 5 half-lives or 1 week, whichever is longer, before baseline [Day -1]) be receiving oral antipsychotic medications; monoamine oxidase inhibitors; anticonvulsants (eg, lamotrigine, Depakote); tricyclic antidepressants (eg, imipramine, desipramine); selective serotonin reuptake inhibitors; or any other psychoactive medications except for as needed anxiolytics (eg, lorazepam, chloral hydrate).
10. Pregnant, lactating, or less than 3 months postpartum.
11. If, in the opinion of the investigator (and/or Sponsor), subject is unsuitable for enrollment in the study or subject has any finding that, in the view of the investigator (and/or Sponsor), may compromise the safety of the subject or affect his/her ability to adhere to the protocol visit schedule or fulfill visit requirements.
12. Positive test for coronavirus (COVID-19) within 2 weeks before screening and at screening.
13. Subjects with extreme concerns relating to global pandemics, such as COVID-19, that preclude study participation.
14. Subject has had psychiatric hospitalization(s) for more than 30 days (cumulative) during the 90 days before screening.
15. Subject has a history of treatment resistance to schizophrenia medications defined as failure to respond to 2 adequate courses of pharmacotherapy (a minimum of 4 weeks at an adequate dose per the label) or required clozapine within the last 12 months.
16. Subjects with prior exposure to KarXT.
17. Subjects who experienced any adverse effects due to xanomeline or trospium.
18. Participation in another clinical study in which the subject received an experimental or investigational drug agent within 3 months before screening.
19. Risk of violent or destructive behavior.
20. Current involuntary hospitalization or incarceration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inder Kaul, MD, Study Director — Karuna Therapeutics
Locations (32):
- United States (20):
  - Pillar Clinical Research, Bentonville, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - Clinical Innovations, Inc, Bellflower, California
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Research, LLC., Garden Grove, California
  - CNS Network, Long Beach, California
  - NRC Research Institute, Orange, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Behavioral Clinical Research, Inc., Hollywood, Florida
  - Larkin Behavioral Health Services, Hollywood, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - AMITA Health Center for Psychiatric Research, Chicago, Illinois
  - Uptown Research Institute, Chicago, Illinois
  - AMITA Health Center for Psychiatric Research, Hoffman Estates, Illinois
  - Hassman Research Institute, Berlin, New Jersey
  - Hassman Research Institute, Marlton, New Jersey
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
- Ukraine (12):
  - Dnipropetrovsk Regional Clinical Hospital named after I.I. Mechnikov, Dnipro
  - Institute of Neurology, Psychiatry and Narcology of the National Academy of Medical Sciences of Ukraine, Kharkiv
  - Regional Clinical Psychiatric Hospital No. 3, Adult Psychiatric Department No. 3, Kharkiv
  - Regional Clinical Psychiatric Hospital No. 3, Psychiatric Department for First Episode Psychosis, Kharkiv
  - Kherson Regional Institution of Mental Care, Kherson
  - Kyiv City Psychoneurological Hospital #2, Kyiv
  - Kyiv Regional Medical Incorporation "Psychiatry", Center for Novel Treatment and Rehabilitation of Psychotic Disorders, Kyiv
  - Lviv Regional Clinical Psychiatric Hospital, Department #20, Lviv
  - Lviv Regional Clinical Psychiatric Hospital, Department #25, Lviv
  - Regional Institution of Mental Psychiatric Care of the Poltava Regional Council, Poltava
  - Cherkasy Regional Psychiatric Hospital of Cherkasy Regional Council, Smila
  - M.I. Pyrogov Vinnytsya National Medical University, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung PP, Breier A, Zhu H, Kaul I, Marcus RN. Xanomeline and Trospium Chloride for the Treatment of Agitation Associated With Schizophrenia: PANSS-Excited Component Results From 3 Randomized, Double-Blind, Placebo-Controlled EMERGENT Trials. J Clin Psychiatry. 2025 Mar 24;86(2):24m15668. doi: 10.4088/JCP.24m15668. PMID 40215379
- [Derived] Citrome L, Neugebauer NM, Meli AA, Kando J. Xanomeline and Trospium Chloride Versus Placebo for the Treatment of Schizophrenia: A Post Hoc Analysis of Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. Neuropsychiatr Dis Treat. 2025 Apr 5;21:761-773. doi: 10.2147/NDT.S503494. eCollection 2025. PMID 40212458
- [Derived] Kaul I, Claxton A, Sawchak S, Sauder C, Brannan SK, Raj E, Ruan S, Konis G, Brown D, Cutler AJ, Marcus R. Safety and Tolerability of Xanomeline and Trospium Chloride in Schizophrenia: Pooled Results From the 5-Week, Randomized, Double-Blind, Placebo-Controlled EMERGENT Trials. J Clin Psychiatry. 2025 Feb 26;86(1):24m15497. doi: 10.4088/JCP.24m15497. PMID 40047530
- [Derived] Kaul I, Sawchak S, Walling DP, Tamminga CA, Breier A, Zhu H, Miller AC, Paul SM, Brannan SK. Efficacy and Safety of Xanomeline-Trospium Chloride in Schizophrenia: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Aug 1;81(8):749-756. doi: 10.1001/jamapsychiatry.2024.0785. PMID 38691387

RESULTS

PARTICIPANT FLOW:
Groups:
- KarXT: All participants assigned to KarXT started on a lead-in dose of KarXT 50/20 (xanomeline 50 mg/trospium chloride 20 mg) BID for the first 2 days (Days 1 and 2) followed by KarXT 100/20 (xanomeline 100 mg/trospium chloride 20 mg) BID for the remainder of Week 1 (Days 3 to 7). At Visit 5 (Day 8), dosing was to be titrated upwards to KarXT 125/30 BID unless the participant experienced AEs from the previous dose of KarXT 100/20 BID. All participants who were increased to KarXT 125/30 BID, depending on clinical response and tolerability, had the option to return to KarXT 100/20 BID for the remainder of the treatment period.
- Placebo: Participants received matching oral placebo treatment twice per day
Period: Overall Study
Arm/Group | KarXT | Placebo
Started (Started=Randomized) | 125 | 131
Recieved Treatment | 125 | 128
Completed | 79 | 93
Not Completed | 46 | 38
Not completed — Changes in condition making participant ineligible for further treatment | 1 | 0
Not completed — Progressive Disease | 0 | 4
Not completed — Adverse Event | 8 | 7
Not completed — Other Reasons | 0 | 1
Not completed — Suicidal or assaultive behavior | 0 | 2
Not completed — Protocol Violation | 2 | 2
Not completed — Consent Withdrawn | 35 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KarXT | Placebo | Total
Number analyzed (Participants) | 125 | 131 | 256
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (11.44) | 42.6 (12.19) | 43.1 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 27 | 65
  Male | 87 | 104 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 14 | 32
  Not Hispanic or Latino | 107 | 117 | 224
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 79 | 77 | 156
  White | 45 | 53 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 5
Description: The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of participants with schizophrenia and is widely used in the study of antipsychotic therapy. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. The positive symptoms in schizophrenia are the excess or distortion of normal function such as hallucinations, delusions, grandiosity, and hostility, and the negative symptoms in schizophrenia are the diminution or loss of normal functions. PANSS total score is the sum of all 30 items with a minimum score of 30 and a maximum score of 210. Higher scores indicate more severe symptoms. The PANSS Total Score is then the sum of the positive, negative, and general psychopathology symptom scores. Baseline is defined as the PANSS score at screening.
Time Frame: From baseline up to Week 5
Population: All participants who were randomized, received at least 1 dose of study drug, had a baseline PANSS assessment, and had at least 1 post-baseline PANSS assessment
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 114 | 120
Score on a scale | -20.6 (1.584) | -12.2 (1.552)

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Positive Score at Week 5
Description: PANSS positive score is the sum of all PANSS 7 positive symptom scales with a minimum score of 7 and a maximum score of 49. Higher scores indicate more severe symptoms. Participants are rated from 1 to 7 on each symptom scale. The positive symptoms in schizophrenia are the excess or distortion of normal function such as hallucinations, delusions, grandiosity, and hostility. If a patient has a PANSS assessment recorded and no more than 2 items are missing from the PANSS positive scales, then the PANSS Positive Score will be calculated as the average of the non-missing items multiplied by 7. If 3 or more items are missing (> 30%) at a particular visit, the respective positive score at the visit will not be calculated and will be treated as missing data. Baseline is defined as the PANSS score at screening.
Time Frame: From baseline up to Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 114 | 120
Score on a scale | -7.1 (0.499) | -3.6 (0.492)

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Negative Score at Week 5
Description: PANSS negative score is the sum of all PANSS 7 negative symptom scales with a minimum score of 7 and a maximum score of 49. Higher scores indicate more severe symptoms. Participants are rated from 1 to 7 on each symptom scale. The negative symptoms in schizophrenia are the diminution or loss of normal functions. If a participant has a PANSS assessment recorded, and no more than 2 items are missing from the PANSS negative scales, then the PANSS Negative Score will be calculated as the average of the non-missing items multiplied by 7. If 3 or more items are missing (> 30%) at a particular visit, the respective negative score at the visit will not be calculated and will be treated as missing data. Baseline is defined as the PANSS score at screening.
Time Frame: From baseline up to Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 114 | 120
Score on a scale | -2.7 (0.412) | -1.8 (0.405)

4. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Negative Marder Factor Score Change From Baseline at Week 5
Description: PANSS Marder factor score is the sum of 5 negative scales and 2 general scales (N1. Blunted affect; N2. Emotional withdrawal; N3. Poor rapport; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity; G7. Motor retardation; and G16. Active social avoidance). Participants are rated from 1 to 7 on each symptom scale. Higher score indicates more severe symptoms. The negative symptoms in schizophrenia are the diminution or loss of normal functions. Baseline is defined as the PANSS score at screening.
Time Frame: From baseline up to Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 114 | 120
Score on a scale | -3.5 (0.484) | -2.7 (0.475)

5. Secondary Outcome: Clinical Global Impression-Severity (CGI-S) Score Change From Baseline at Week 5
Description: Clinical Global Impression-Severity (CGI-S) Score is a measurement to evaluate severity and treatment response in schizophrenia. Completed independently by a clinician, the CGI-S assesses extremely ill patients, by asking 1 question and providing a rating based upon observed and reported symptoms, behavior, and function in the past 7 days to reflect the average severity level across the 7 days. Higher score indicates more severe illness. The CGI-S categorizes the severity of the illness as: 1 = Normal, not at all ill; 2 = Borderline mentally ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; and 7 = Among the most extremely ill patients. This scale reflects the total score. Baseline is defined as CGI-S score at screening. The change from baseline in total score is reported.
Time Frame: From baseline up to Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 114 | 120
Score on a scale | -1.1 (0.091) | -0.6 (0.088)

6. Secondary Outcome: Number of Participants Who Achieve >=30% Reduction in Positive and Negative Symptoms Scale (PANSS) Total Score From Baseline to Week 5
Description: Positive and Negative Syndrome Scale (PANSS) is a scale used for measuring symptom severity of subjects with schizophrenia and is widely used in the study of antipsychotic therapy. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Subjects are rated from 1 to 7 on each symptom scale. The positive symptoms in schizophrenia are the excess or distortion of normal function such as hallucinations, delusions, grandiosity, and hostility, and the negative symptoms in schizophrenia are the diminution or loss of normal functions. PANSS total score is the sum of all 30 items with a minimum score of 30 and a maximum score of 210. Higher scores indicate more severe symptoms. The PANSS Total Score is then the sum of the positive, negative, and general psychopathology symptom scores. Baseline is defined as screening.
  Note: Floor adjusted data were used for this analysis. Floor adjusted total score = total score - 30.
Time Frame: From baseline up to Week 5
Population: All participants who were randomized, received at least 1 dose of study drug, had a baseline PANSS assessment, and had at least 1 post-baseline PANSS assessment, and had a PANSS score at Week 5
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 79 | 91
Participants | 40 | 23

7. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to Day 42
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 125 | 128
Participants | 88 | 64

8. Secondary Outcome: Number of Participants Experiencing Cholinergic Symptom Adverse Event
Description: The number of participants experiencing adverse events related to procholinergic symptoms (believed to be associated with xanomeline) and anticholinergic symptoms (believed to be associated with trospium) symptoms. Examples of procholinergic symptoms include vomiting, nausea, diarrhea, sweating and hyper-salivation. Examples of anticholinergic include dizziness, confusion, hallucinations, and somnolence.
Time Frame: From first dose up to Day 42
Population: All participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 125 | 128
Participants
  At Least One Procholinergic Symptom Adverse Event | 38 | 3
  At Least One Anticholinergic Symptom Adverse Event | 33 | 8

9. Secondary Outcome: Change From Baseline in Simpson-Angus Scale Total Score (SAS)
Description: The Simpson-Angus Scale (SAS) is an established instrument to measure drug-related extrapyramidal syndromes. It is a 10-item testing instrument used to assess gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, glabella tap, tremor, and salivation. The range of scores is from 0 to 40 with increased scores indicating increased severity. Baseline is defined as the Simpson-Angus Scale score recorded on Day -1.
Time Frame: From baseline up to week 5
Population: All treated participants
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 125 | 128
Score on a Scale | -0.1 (0.56) | -0.1 (0.36)

10. Secondary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS) Total Score
Description: The BARS for akathisia is a rating scale used to assess the severity of drug-induced akathisia, or restlessness, involuntary movements and inability to sit still. The range of scores is 0 to 14, with higher scores indicating greater severity. Baseline is defined as the BARS score recorded on Day -1.
Time Frame: From baseline up to week 5
Population: All treated participants with evaluable BARS total score at the prespecified timepoint
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 79 | 91
Score on a Scale | -0.1 (0.75) | -0.1 (0.88)

11. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score
Description: The AIMS is a rating scale that is used to measure involuntary movements known as tardive dyskinesia, which can sometimes develop as a side effect of long-term treatment with antipsychotic medications. This measurement was a 12-item scale to assess orofacial, extremity, and truncal movements as well as the overall severity, incapacitation, and the participant's level of awareness of the movements. Items are scored from 0 (none) to 4 (severe). A higher score indicates more severe dyskinesia. Baseline is defined as the AIMS score recorded on Day -1. The total score is the sum of sub scores for items 1-7. The first 7 items are used to measure the severity of abnormal movements in the orofacial region (4 items: facial muscles, lips, jaw, tongue), upper extremities (1 item), lower extremities (1 item), and trunk (1 item). Change from baseline for the total scores are reported.
Time Frame: From baseline up to week 5
Population: All treated participants with evaluable AIMS total score at the prespecified timepoint
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 79 | 91
Units on a Scale | 0.0 (0.45) | 0.0 (0.15)

12. Secondary Outcome: Number of Participants Who Experienced Weight Change
Description: The number of participants who lost weight, maintained their weight, or gained weight between baseline and week 5. Baseline is defined as measurements taken at screening.
Time Frame: From baseline up to week 5
Population: All treated participants with evaluable weight values at the prespecified timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 78 | 92
Participants
  Lost Weight | 1 | 0
  Maintained Weight1 | 72 | 80
  Gained Weight | 5 | 12

13. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: The change in Body Mass Index (BMI) from baseline up to week 5. BMI is a person's weight in kilograms divided by the square of height in meters. Baseline is defined as measurements taken at screening.
Time Frame: From baseline up to week 5
Population: All treated participants with evaluable BMI values at the prespecified timepoint
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 78 | 92
kg/m^2 | 0.457 (1.1340) | 0.666 (0.570)

14. Secondary Outcome: Change From Baseline in Waist Circumference
Description: The change in waist circumference in centimeters from baseline up to week 5. Baseline is defined as measurements taken at screening.
Time Frame: From baseline up to week 5
Population: All treated participants with evaluable waist circumference values at the prespecified timepoint
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 78 | 92
Centimeters | 1.666 (4.8915) | 1.697 (4.8577)

15. Secondary Outcome: Change From Baseline in Orthostatic Vital Signs - Blood Pressure
Description: The change from baseline in orthostatic diastolic and systolic blood pressure measured while supine and standing after 2 minutes. Baseline is defined as measurements taken at screening.
Time Frame: From baseline up to week 5
Population: All treated participants with evaluable blood pressure values at the prespecified timepoint
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 79 | 92
mmHg
  Supine Systolic Blood Pressure | 1.9 (13.07) | 0.4 (13.00)
  Supine Diastolic Blood Pressure | 2.2 (10.33) | 0.4 (9.30)
  Standing Systolic Blood Pressure | 2.3 (14.07) | 0.1 (12.54)
  Standing Diastolic Blood Pressure | 2.7 (9.93) | 0.1 (8.62)

16. Secondary Outcome: Change From Baseline in Orthostatic Vital Signs - Heart Rate
Description: The change from baseline in orthostatic heart rate measured while supine and standing after 2 minutes. Baseline is defined as measurements taken at screening.
Time Frame: From baseline up to week 5
Population: All treated participants with evaluable heart rate values at the prespecified timepoint
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 79 | 92
beats/min
  Supine Heart Rate | 11.9 (15.72) | 6.1 (14.02)
  Standing Heart Rate | 9.86 (16.58) | 5.8 (13.85)

17. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Mean Heart Rate
Description: The change from baseline up to Day 35 or early termination in ECG mean heart rate. Baseline is defined as measurements taken at screening.
Time Frame: From baseline up to Day 35 or early termination
Population: All treated participants
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 125 | 128
beats/min | 11.5 (14.94) | 6.1 (14.62)

18. Secondary Outcome: Number of Participants Experiencing Clinically Significant Abnormal Physical Examination Results
Description: The number of participants experiencing clinically significant abnormal physical examination results. Baseline is defined as measurements taken at screening.
Time Frame: From baseline up to week 5
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 125 | 128
Participants
  General Appearance - Baseline: number analyzed (Participants) | 123 | 128
  General Appearance - Baseline | 0 | 1
  General Appearance - Day 35: number analyzed (Participants) | 79 | 93
  General Appearance - Day 35 | 0 | 0
  Head, Eyes, Ears, Nose, Throat - Baseline: number analyzed (Participants) | 123 | 128
  Head, Eyes, Ears, Nose, Throat - Baseline | 0 | 0
  Head, Eyes, Ears, Nose, Throat - Day 35: number analyzed (Participants) | 79 | 93
  Head, Eyes, Ears, Nose, Throat - Day 35 | 0 | 0
  Thorax - Baseline: number analyzed (Participants) | 124 | 128
  Thorax - Baseline | 0 | 0
  Thorax - Day 35: number analyzed (Participants) | 79 | 93
  Thorax - Day 35 | 0 | 0
  Abdomen - Baseline: number analyzed (Participants) | 124 | 128
  Abdomen - Baseline | 1 | 0
  Abdomen - Day 35: number analyzed (Participants) | 79 | 93
  Abdomen - Day 35 | 0 | 0
  Cardiac - Baseline: number analyzed (Participants) | 124 | 128
  Cardiac - Baseline | 1 | 0
  Cardiac - Day 35: number analyzed (Participants) | 79 | 93
  Cardiac - Day 35 | 0 | 0
  Musculoskeletal - Baseline: number analyzed (Participants) | 124 | 128
  Musculoskeletal - Baseline | 0 | 0
  Musculoskeletal - Day 35: number analyzed (Participants) | 79 | 93
  Musculoskeletal - Day 35 | 0 | 0
  Circulatory System - Baseline: number analyzed (Participants) | 124 | 128
  Circulatory System - Baseline | 0 | 0
  Circulatory System - Day 35: number analyzed (Participants) | 79 | 93
  Circulatory System - Day 35 | 0 | 0
  Lymphadenopathy - Baseline: number analyzed (Participants) | 124 | 128
  Lymphadenopathy - Baseline | 0 | 0
  Lymphadenopathy - Day 35: number analyzed (Participants) | 79 | 93
  Lymphadenopathy - Day 35 | 0 | 0
  Limited Neurological Examination - Baseline: number analyzed (Participants) | 124 | 128
  Limited Neurological Examination - Baseline | 1 | 0
  Limited Neurological Examination - Day 35: number analyzed (Participants) | 79 | 93
  Limited Neurological Examination - Day 35 | 0 | 0

19. Secondary Outcome: Number of Participants Experiencing Each Suicidal Ideation Scale Category as Per Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS assesses suicidal behavior and ideation on a scale with 4 general categories: suicidal ideation, intensity of ideation, suicidal behavior, and actual attempts. C-SSRS comprehensively identifies suicidal events while limiting the over identification of suicidal behavior. The C-SSRS was administered by a trained rater at the site.
  This study used 2 versions of the C-SSRS. At the Screening Visit, the "Lifetime" version was completed; for all subsequent visits, the "Since Last Visit" version of the C-SSRS was administered.
  Risk for suicidal behavior during the study was determined by the investigator's clinical assessment and C-SSRS as confirmed by the following:
  * Answering "Yes" on items 4 or 5 (C-SSRS - ideation) with the most recent episode occurring within the 2 months before screening, or
  * Answering "Yes" to any of the 5 items (C-SSRS behavior) with an episode occurring within the 12 months before screening. Non-suicidal, self-injurious behavior is not exclusionary.
Time Frame: From screening up to Day 42
Population: All participants who had evaluable C-SSRS data.
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 125 | 120
Participants
  Suicidal Ideation: Participant Wished to be Dead | 1 | 3
  Suicidal Ideation: Non-Specific Active Suicidal Thoughts | 1 | 1
  Suicidal Ideation: Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act | 0 | 1
  Most Severe Ideation Level 1. Least Severe | 0 | 2
  Most Severe Ideation Level 2 | 1 | 0
  Most Severe Ideation Level 3 | 0 | 1
  Intensity of Ideation (Frequency) - Less than once a week | 0 | 1
  Intensity of Ideation (Frequency) - Once a week | 0 | 1
  Intensity of Ideation (Frequency) - 2-5 times a week | 1 | 1
  Intensity of Ideation (Duration) - Fleeting, a few seconds or minutes | 1 | 3
  Controllability - Easily able to control thoughts | 0 | 3
  Controllability - Can control thoughts with little difficulty | 1 | 0
  Deterrents - Does not apply | 0 | 1
  Deterrents - Deterrents definitely stopped participant from attempting suicide | 1 | 2
  Reasons for Ideation - Does not apply | 0 | 2
  Reasons for Ideation - Mostly to end or stop the pain | 0 | 1
  Reasons for Ideation - Completely to end or stop the pain | 1 | 0

20. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC)
Description: AUC is the total area under the plasma drug concentration-time curve from time zero to 12 hours after drug administration. Dose level 125/30 BID at Week 4 (Visit 8 [Day 28]) is reported.
Time Frame: At days 8 and 28
Population: All participants who received at least 1 dose of active study drug and have at least 1 measurable (AUC) plasma concentration of study drug.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 77 | 0
h*pg/mL
  Trospium | 27800 (26000) |
  Xanomeline: number analyzed (Participants) | 76 | 0
  Xanomeline | 50200 (37900) |

21. Secondary Outcome: Maximum Concentration (Cmax)
Description: Cmax is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered and before the administration of a second dose. Dose level 125/30 BID at Week 4 (Visit 8 [Day 28]) is reported.
Time Frame: At days 8 and 28
Population: All participants who received at least 1 dose of active study drug and have at least 1 measurable (Cmax) plasma concentration of study drug.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 79 | 0
pg/mL
  Trospium | 6070 (7780) |
  Xanomeline | 9660 (10500) |

22. Secondary Outcome: Time to Maximum Concentration (Tmax)
Description: Tmax is defined as the time it takes for a drug to reach the maximum concentration (Cmax) after administration of a drug. Dose level 125/30 BID at Week 4 (Visit 8 [Day 28]) is reported.
Time Frame: At days 8 and 28
Population: a. All participants who received at least 1 dose of active study drug and have at least 1 measurable (Tmax) plasma concentration of study drug.
Measure: Median (Full Range); unit: Hours
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 79 | 0
Hours
  Trospium | 1.00 [0.00 to 3.95] |
  Xanomeline | 2.00 [0.00 to 12.00] |

23. Secondary Outcome: Mean Observed Hemoglobin Levels
Description: The mean observed Hemoglobin levels are displayed as measured at the specified timepoints. Baseline is defined as first dose.
  Reference Range:
  Male: 138 - 172 g/L Female: 121 - 151 g/L
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable hemoglobin levels at the specified timepoint
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 124 | 127
g/L
  Baseline | 142.30 (18.098) | 142.71 (15.166)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 88 | 97
  Week 3 (Visit 7 [Day 21]) | 144.54 (19.096) | 146.27 (14.335)
  Week 5 (Visit 10 [Day 35])/Early-Termination: number analyzed (Participants) | 104 | 110
  Week 5 (Visit 10 [Day 35])/Early-Termination | 142.94 (19.175) | 144.40 (15.416)

24. Secondary Outcome: Mean Observed Hematocrit Levels
Description: The mean observed Hematocrit levels are displayed in percentages as measured at the specified timepoints. Baseline is defined as first dose.
  Reference Range:
  Male: 40.7 - 50.3% Female: 36.1 - 44.3%
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable hematocrit levels at the specified timepoint
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 124 | 127
Percentage
  Baseline | 44.52 (5.232) | 44.51 (4.553)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 87 | 96
  Week 3 (Visit 7 [Day 21]) | 45.12 (5.416) | 45.25 (4.306)
  Week 5 (Visit 10 [Day 35])/Early-Termination: number analyzed (Participants) | 102 | 109
  Week 5 (Visit 10 [Day 35])/Early-Termination | 44.51 (5.491) | 44.71 (4.595)

25. Secondary Outcome: Mean Observed Erythrocyte Levels
Description: The mean observed erythrocyte levels are displayed as measured at the specified timepoints. Baseline is defined as first dose.
  Reference Range:
  Male: 4.7 - 6.1 10^12 cells/L Female: 4.2 - 5.4 10^12 cells/L
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable erythrocyte levels at the specified timepoint
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 124 | 127
10^12 cells/L
  Baseline | 5.025 (0.5072) | 4.894 (0.4498)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 88 | 97
  Week 3 (Visit 7 [Day 21]) | 5.130 (0.4986) | 5.165 (1.2161)
  Week 5 (Visit 10 [Day 35])/Early-Termination: number analyzed (Participants) | 104 | 110
  Week 5 (Visit 10 [Day 35])/Early-Termination | 5.058 (0.5339) | 5.003 (0.5139)

26. Secondary Outcome: Mean Observed Platelets Levels
Description: The mean observed platelet levels are displayed as measured at the specified timepoints. Baseline is defined as first dose.
  Reference Range:
  150-450 10^9 cells/L
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable platelet levels at the specified timepoint
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 124 | 127
10^9 cells/L
  Baseline | 334.04 (96.465) | 328.65 (92.288)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 88 | 97
  Week 3 (Visit 7 [Day 21]) | 334.47 (80.273) | 320.21 (73.757)
  Week 5 (Visit 10 [Day 35])/Early-Termination: number analyzed (Participants) | 104 | 110
  Week 5 (Visit 10 [Day 35])/Early-Termination | 336.59 (88.455) | 327.91 (75.834)

27. Secondary Outcome: Mean Observed Leukocytes Levels
Description: The mean observed leukocytes levels are displayed as measured at the specified timepoints. Baseline is defined as first dose.
  Reference Range:
  4.5-10 10^9 cells/L
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable leukocytes levels at the specified timepoint
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 124 | 127
10^9 cells/L
  Baseline | 5.971 (1.9465) | 6.384 (2.1421)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 88 | 97
  Week 3 (Visit 7 [Day 21]) | 6.046 (1.8090) | 6.252 (1.6685)
  Week 5 (Visit 10 [Day 35])/Early-Termination: number analyzed (Participants) | 104 | 110
  Week 5 (Visit 10 [Day 35])/Early-Termination | 6.199 (2.1814) | 6.184 (1.7208)

28. Secondary Outcome: Mean Observed Lymphocytes Levels
Description: The mean observed lymphocytes levels are displayed as measured at the specified timepoints. Baseline is defined as first dose.
  Reference Range:
  1-4.8 10^9 cells/L
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable lymphocytes levels at the specified timepoint
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 124 | 127
10^9 cells/L
  Baseline | 2.749 (0.9408) | 3.094 (3.9283)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 87 | 93
  Week 3 (Visit 7 [Day 21]) | 2.834 (0.9890) | 2.976 (0.9431)
  Week 5 (Visit 10 [Day 35])/Early-Termination: number analyzed (Participants) | 101 | 105
  Week 5 (Visit 10 [Day 35])/Early-Termination | 3.000 (1.2748) | 2.792 (0.8456)

29. Secondary Outcome: Mean Observed Activated Partial Thromboplastin Time
Description: The mean observed activated partial thromboplastin times in seconds are displayed as measured at the specified timepoints. Baseline is defined as first dose.
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable activated partial thromboplastin time data at the specified timepoint
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 124 | 127
Seconds
  Baseline | 30.75 (4.412) | 31.75 (5.897)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 85 | 90
  Week 3 (Visit 7 [Day 21]) | 32.43 (4.798) | 33.55 (7.858)
  Week 5 (Visit 10 [Day 35])/Early-Termination: number analyzed (Participants) | 99 | 103
  Week 5 (Visit 10 [Day 35])/Early-Termination | 31.48 (3.636) | 33.04 (6.775)

30. Secondary Outcome: Mean Observed Prothrombin Time
Description: The mean observed prothrombin times are displayed as measured at the specified timepoints. Baseline is defined as first dose.
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable prothrombin time data at the specified timepoint
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 123 | 126
Seconds
  Baseline | 1.00 (0.091) | 1.01 (0.086)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 86 | 88
  Week 3 (Visit 7 [Day 21]) | 1.02 (0.096) | 1.00 (0.086)
  Week 5 (Visit 10 [Day 35])/Early-Termination: number analyzed (Participants) | 99 | 102
  Week 5 (Visit 10 [Day 35])/Early-Termination | 1.01 (0.078) | 1.00 (0.083)

31. Secondary Outcome: Mean Observed Urinalysis - pH
Description: The mean observed pH of participants' urine are displayed as measured at the specified timepoints. Baseline is defined as first dose. Urinalysis was completed using dipstick. Urinalysis was not completed if the local dipstick was normal.
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable urine pH data at the specified timepoint
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 89 | 82
pH
  Baseline | 5.52 (0.676) | 5.59 (0.800)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 57 | 59
  Week 3 (Visit 7 [Day 21]) | 5.33 (0.476) | 5.48 (0.748)
  Week 5 (Visit 10 [Day 35]/Early Termination): number analyzed (Participants) | 56 | 59
  Week 5 (Visit 10 [Day 35]/Early Termination) | 5.48 (0.687) | 5.45 (0.621)

32. Secondary Outcome: Mean Observed Urinalysis - Prolactin
Description: The mean observed prolactin levels of participants' urine are displayed as measured at the specified timepoints. Baseline is defined as first dose. Urinalysis was not completed if the local dipstick was normal.
Time Frame: From baseline up to Days 21, 35, or early temination
Population: All treated participants with evaluable urine prolactin data at the specified timepoints
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 125 | 122
ug/L
  Baseline | 18.08 (21.767) | 17.38 (21.920)
  Week 3 (Visit 7 [Day 21]): number analyzed (Participants) | 88 | 90
  Week 3 (Visit 7 [Day 21]) | 17.49 (19.422) | 14.50 (12.064)
  Week 5 (Visit 10 [Day 35]/Early Termination): number analyzed (Participants) | 102 | 105
  Week 5 (Visit 10 [Day 35]/Early Termination) | 19.46 (24.668) | 15.56 (13.463)

33. Secondary Outcome: The Number of Participants With Positive Drug Screen Results
Description: A National Institute on Drug Abuse-5 urine drug screen (cannabinoids or marijuana, phencyclidine, amphetamines, opiates, and cocaine) was performed at screening and at baseline (Visit 2a [Day -1]). If a participant left the study site, they were to have a urine drug screen and test for alcohol (breathalyzer or urine alcohol level) upon returning to the study site.
Time Frame: At screening, at Dat -1, and upon return from departure from study site at any time up to Day 42
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 125 | 128
Participants | 3 | 1

34. Secondary Outcome: The Number of Participants With Elevated Liver Function Test Results
Description: The liver function test results (ALT, AST, ALP, total bilirubin, GGT) were specifically monitored to watch for any participants who met the FDA drug-induced liver injury (DILI) criteria. A summary of elevated liver function test results by visit is provided. Baseline is defined as measurements taken at screening.
  Monitoring for DILI criteria includes close observation initiated with ALT or AST >3 × ULN; discontinuation of treatment should be considered if ALT or AST >8 × ULN, ALT or AST >5 × ULN for more than 2 weeks, ALT or AST >3 × ULN and (total bilirubin >2 × ULN or international normalized ratio >1.5), or ALT or AST >3 × ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia (>5%).
Time Frame: From screening up to Day 42
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 125 | 128
Participants
  Baseline - Bilirubin (umol/L) > 1. 5 x ULN | 1 | 0
  Baseline - Gamma Glutamyl Transferase (U/L) > 2 x ULN | 4 | 4
  Baseline - Alanine Aminotransferase (U/L) > 3 x ULN | 0 | 0
  Baseline - Aspartate Aminotransferase (U/L) > 3 x ULN | 0 | 0
  Baseline - Alkaline Phosphatase (U/L) > 105 x ULN | 0 | 0
  Baseline - Hy's Law Cases | 0 | 0
  Visit 4 Day 7 - Gamma Glutamyl Transferase (U/L) > 2 x ULN | 0 | 1
  Visit 7 Day 21 - Alanine Aminotransferase (U/L) > 3 x ULN | 1 | 0
  Visit 7 Day 21 - Alanine Aminotransferase (U/L) > 5 x ULN | 2 | 0
  Visit 7 Day 21 - Aspartate Aminotransferase (U/L) > 3 x ULN | 1 | 0
  Visit 7 Day 21 - Alkaline Phosphatase (U/L) > 2 x ULN | 1 | 0
  Visit 7 Day 21 - Gamma Glutamyl Transferase (U/L) > 2 x ULN | 6 | 1
  Visit 10 Day 35 - Alanine Aminotransferase (U/L) > 3 x ULN | 0 | 1
  Visit 10 Day 35 - Alanine Aminotransferase (U/L) > 5 x ULN | 1 | 0
  Visit 10 Day 35 - Alkaline Phosphatase (U/L) > 1. 5 x ULN | 1 | 0
  Visit 10 Day 35 - Gamma Glutamyl Transferase (U/L) > 2 x ULN | 4 | 1
  Visit 10 or Early Termination Alanine Aminotransferase (U/L) >3x ULN | 0 | 1
  Visit 10 or Early Termination - Alanine Aminotransferase (U/L) >5x ULN | 1 | 0
  Visit 10 or Early Termination - Alkaline Phosphatase (U/L) > 1. 5 x ULN | 1 | 1
  Visit 10 or Early Termination - Bilirubin (umol/L) > 2 x ULN | 1 | 0
  Visit 10 or Early Termination - Gamma Glutamyl Transferase (U/L) > 2 x ULN | 7 | 1
  Visit 11 Day 42 - Bilirubin (umol/L) > 1. 5 x ULN | 1 | 0
  Visit 11 Day 42 - Gamma Glutamyl Transferase (U/L) > 2 x ULN | 3 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 20 months). SAEs and Other AEs were assessed from first dose up to Day 42.
Arm/Group | KarXT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/131
Serious Adverse Events (participants affected / at risk) | 1/125 | 0/128
Other Adverse Events (participants affected / at risk) | 69/125 | 36/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT (N=125) | Placebo (N=128)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT (N=125) | Placebo (N=128)
Constipation (Gastrointestinal disorders) | 16 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Dyspepsia (Gastrointestinal disorders) | 20 | 2
Nausea (Gastrointestinal disorders) | 24 | 2
Vomiting (Gastrointestinal disorders) | 20 | 1
Headache (Nervous system disorders) | 14 | 15
Anxiety (Psychiatric disorders) | 2 | 8
Insomnia (Psychiatric disorders) | 7 | 10
Hypertension (Vascular disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT04738123/Prot_SAP_000.pdf